CLINICAL TRIAL: NCT01968161
Title: An Open-label Switch Study to Asenapine in the Early Stage of Psychosis
Brief Title: Investigator Initiated Study - Asenapine Early Psychosis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centre de Recherche de l'Institut Universitaire en Santé Mentale de Québec (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIS - Switch Asenapine
Record Dates: First submitted 2013-10-16; First posted 2013-10-23 (Estimated); Last update posted 2014-01-09 (Estimated); Status verified 2014-01

CONDITIONS: Schizophrenia and Disorders With Psychotic Features; Disorders
MeSH Terms: conditions — Schizophrenia Spectrum and Other Psychotic Disorders; Disease | interventions — asenapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Asenapine (Other): Open label switch to asenapine: asenapine will be introduced at the target dose (5 mg bid)
  Interventions: Drug: Asenapine

INTERVENTIONS:
Drug: Asenapine

SUMMARY:
We propose a use of a unique facility, the databank at the CNDV, to examine the impact of switching subjects to asenapine in an open-label naturalistic setting. This offers the following advantages: i) providing data on a particularly important population, i.e., subjects who are at the inception of treatment for a psychotic disorder and who are likely to remain on a given drug on a long-term basis; ii) its inclusion in a rich clinical setting, with a clinical team dedicated to provide innovative interventions; iii) its naturalistic design, that will allow to obtain data that will be applicable to "real-life" clinical settings; indeed, subjects who will be switched to asenapine within the current project are those we would switch to this drug in our daily practice.

ELIGIBILITY:
Inclusion Criteria:

* Meeting DSM-IV criteria for schizophrenia (SZ) or related SZ spectrum psychotic disorders
* having provided a consent to include data on our databank,and being able to provide informed consent
* willingness to participate to the assessments
* being over 18 years of age
* being in a clinical situation that warrants switch to asenapine

Exclusion Criteria:

* suffering from a primary drug-induced psychosis
* being at significant risk for suicide or assault
* unstable medical condition
* persistence of psychotic symptoms despite adequate treatment to an extent that clozapine would be required
* being treated with antipsychotic for 5 years or more
* having contraindications(allergy to asenapine)
* being pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2013-10; Primary Completion 2014-02 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Impact of switching to asenapine | 3 months

SECONDARY OUTCOMES:
Predictors of successful switch to asenapine | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Marc-André Roy, MD, Principal Investigator — Centre de Recherche de l'Institut Universitaire en Santé Mentale de Québec
Locations (1):
- Clinique Notre-Dame des Victoires, Québec, Quebec, Canada